CLINICAL TRIAL: NCT04402307
Title: Effect of Training of Patients With Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regionshospital Nordjylland (Other Government)
Responsible Party: Principal Investigator, Dorte Melgaard Kristiansen, Seniorresearcher, research coordinator, ph.d., Regionshospital Nordjylland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RHN_DMK_05
Record Dates: First submitted 2019-04-01; First posted 2020-05-26 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Dysphagia
Keywords: Training; Effect; Elderly
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Usual care to patients with dysphagia
- Training (Experimental): Chin Tuck Against Resistance to patients with dysphagia
  Interventions: Other: Chin Tuck Against Resistance

INTERVENTIONS:
Other: Chin Tuck Against Resistance — Training in 6 weeks 3 times a day.
  Arms: Training

SUMMARY:
Effect of training of patients with dysphagia

DETAILED DESCRIPTION:
A randomised controlled study in the effect of training in patients with dysphagia.

The patients are randomised for training or for usual care.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with dysphaigia
* Patients living in the participating locations

Exclusion Criteria:

* Patients who are linguistically or cognitively unable to participate
* Patients who are unable to collaborate about the training
* Palliative patients
* Patients with a probe

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Readmission | 6 months
  Number of readmissions within 6 months

SECONDARY OUTCOMES:
Change in Quality of life | 3 months
  Level of quality of life - measured with Dysphagia Handicap Index questionnaire
Cost effectiveness | 6 months
  Economic evaluation of training compared to usual care, measured with EQ-5D
Mortality | 6 months
  Mortality in patients with dysphagia within 6 months
Swallowing function | 3 months
  Aspiration (yes/no) - measured with Volume Viscosity Swallow Test

CONTACTS AND LOCATIONS:
Overall Officials: Dorte M Kristiansen, PhD, Principal Investigator — Regionshospital Nordjylland
Locations (8):
- Denmark (8):
  - Jammerbugt municipality, Brovst
  - Brøndby municipality, Brøndby
  - Frederikshavn municipality, Frederikshavn
  - Hjørring municipality, Hjørring
  - Kolding municipality, Kolding
  - Odense municipality, Odense
  - Slagelse municipality, Slagelse
  - Tønder municipality, Tønder